CLINICAL TRIAL: NCT06343857
Title: Spontaneous Multicenter Prospective Observational Study for the Development of Joint Wellness Self-assessment Forms
Brief Title: Joint Self-Assessment Forms for Knee, Ankle and Shoulder
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Leo Massari, MD, University Hospital of Ferrara
Other Study IDs: CE-AVEC 878/2022/Oss/AOUFe
Record Dates: First submitted 2024-03-19; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Anatomical site: Subjects who have requested an orthopaedic specialist examination for the knee, or ankle or shoulder
  Interventions: Diagnostic Test: self-assessment questionnaire

INTERVENTIONS:
Diagnostic Test: self-assessment questionnaire — Completion of the anatomical site-specific self-assessment questionnaire.

SUMMARY:
The present study represents the pilot phase of the project aimed at developing anatomical site-specific self-assessment questionnaires (shoulder, knee and ankle) that can advise the subject of the need for an orthopaedic specialist examination.

The pilot phase of the project involves the collection of data from questionnaires in a population of subjects who have requested an orthopaedic consultation for the anatomical site covered by the questionnaire. Each questionnaire consists of questions designed to collect information about the patient's subjective condition.

The data collected from the questionnaires will be used to evaluate the statistical significance (p value) of each question in the questionnaire in relation to the outcome of the orthopaedic specialist visit. Through a multivariate logistic analysis of the answers given by the subject, it will be possible to 'weight' each answer to obtain a final value that gives an indication of an orthopaedic specialist visit.

DETAILED DESCRIPTION:
With the present study, an initial exploratory phase is conducted aimed at developing anatomical site-specific self-assessment questionnaires (shoulder, knee, and ankle) capable of directing the subject to the need for an orthopedic specialist visit. The questionnaire will allow the subject to understand whether his or her symptomatology indicates the presence of a clinical condition requiring orthopedic specialist examination. In this way, it will be possible to identify patients in need of a specialist visit in a timely manner, avoiding chronicity of the painful symptomatology and allowing early diagnosis and potentially faster functional recovery.

To this end, starting from the analysis of clinically validated 1-10 questionnaires, orthopedic specialists afferent to the University of Ferrara, the Rizzoli Orthopedic Institute, and the Galeazzi Orthopedic Institute collaboratively developed questionnaires with the following characteristics:

1. Subjectivity: the questions in the questionnaires require an answer that reflects a specific condition of the subject, e.g. ability to carry out daily or sporting activities.
2. Specificity: the questions in the questionnaires are specific to the anatomical district (shoulder, knee, ankle).
3. Simplicity: being a questionnaire completed by the subject in complete autonomy, the questions are written in simple language and the compilation method is intuitive.
4. Reliability: the score obtained from completing the questionnaires must be able to distinguish subjects who require further diagnostic tests from subjects who require pharmacological therapy, physical therapy, or no therapy.

The self-assessment forms are provided as an attachment to the clinical protocol.

The present study represents the pilot phase of the project aimed at developing self-assessment questionnaires specific to anatomical site (shoulder, knee, and ankle) and involves the collection of data from self-assessment forms in a population of subjects who have requested an orthopedic specialist visit for the anatomical site covered by the questionnaire. As part of the proposed study, the answers provided by the patient will be compared with the outcome of the orthopedic specialist visit.

The data collected from the questionnaires will be used to: 1. evaluate the statistical significance (p value) of each question in the questionnaire in relation to the result of the orthopedic specialist visit. and 2. assign a score to each response in relation to the outcome of the orthopedic specialist visit.

The proposed study will allow us to develop self-assessment questionnaires which, based on simple questions, can direct the patient towards the need for an orthopedic specialist visit.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have requested an orthopaedic specialist examination for the anatomical site covered by the self-assessment form;
* Age 18 years or older;
* Comprehension of the Italian language.

Exclusion Criteria:

* Surgery within the previous 12 months at the anatomical site covered by the self-assessment form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: outpatients, orthopaedic clinic
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Observation of the distribution of questionnaire responses for each anatomical site. | baseline
  The data collected from the questionnaires will be used to assess the statistical significance (p value) of each question in the questionnaire in relation to the outcome of the orthopedic specialist examination

SECONDARY OUTCOMES:
Therapeutic indication of the orthopaedic specialist for each subject participating in the study | baseline
  The collection of the orthopaedic specialist's opinion on the therapeutic indication for each subject participating in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Leo Massari, MD, Principal Investigator — Azienda Ospedaliera-Universitaria Arcispedale S. Anna di Ferrara
Locations (2):
- Italy (2):
  - IRCCS Istituto Ortopedico Rizzoli, Clinica Ortopedica e Traumatologica II, Bologna, BO
  - Unità Operativa di Chirurgia della Spalla I.R.C.C.S. Ospedale Galeazzi-Sant'Ambrogio, Milan, MI

IPD SHARING:
Plan to Share IPD: Undecided